CLINICAL TRIAL: NCT02809014
Title: In Vivo Evaluation of an Experimental Fluoride-containing Dentifrice With Hydrocolloid
Acronym: FdentifriceT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fabio Correia Sampaio (Other)
Responsible Party: Sponsor-Investigator, Fabio Correia Sampaio, Professor, Federal University of Paraíba
Organization: Federal University of Paraíba (Other)
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: Fluoride dentifrice tara
Record Dates: First submitted 2016-06-17; First posted 2016-06-22 (Estimated); Last update posted 2022-05-20 (Actual); Status verified 2022-05

CONDITIONS: Dental Caries
Keywords: Fluoride; Dental caries; Dentifrice
MeSH Terms: conditions — Dental Caries | interventions — Dentifrices; tara gum

STUDY DESIGN:
Intervention Model Description: The intervention was based on the use of dentifrices: experimental dentifrices: placebo (without F and without tara gum), 100-TGF (NaF associated with tara gum, 1100 mg/L F), 50-TGF (50% NaF associated with tara gum + 50% free NaF, 1100 mg/L F), positive control (PC) (free NaF, 1100 mg/L F), and TG (with tara gum and without F) (Savoy SA, São Paulo, Brazil).
Who Masked: Participant, Care Provider, Investigator
Masking Description: masking by color and QR code
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Placebo (Placebo Comparator): Dentifrice without fluoride and tara gum.
  Interventions: Other: Dentifrice F-Complex; Other: Dentifrice F-Complex + NaF; Other: Dentifrice standard; Other: Dentifrice with tara gum
- Dentifrice standard (Active Comparator): Dentifrice 1100 ppm sodium fluoride (NaF) without tara gum. Positive control
  Interventions: Other: Dentifrice standard
- Dentifrice with tara gum (Placebo Comparator): Dentifrice without fluoride but with hydrocolloid tara gum.
  Interventions: Other: Dentifrice with tara gum
- Dentifrice F-Complex + NaF (Experimental): Dentifrice experimental with fluoride (1100 ppm) being half of fluoride incorporated in tara gum and other half freeform of NaF
  Interventions: Other: Dentifrice F-Complex + NaF
- Dentifrice F-Complex (Experimental): Dentifrice experimental with fluoride (1100 ppm) all incorporated in tara gum.
  Interventions: Other: Dentifrice F-Complex

INTERVENTIONS:
Other: Dentifrice F-Complex — Use of few of dentifrice on brushing for one week, twice day.
  Arms: Dentifrice F-Complex; Placebo
Other: Dentifrice F-Complex + NaF — Use of few of dentifrice on brushing for one week, twice day.
  Arms: Dentifrice F-Complex + NaF; Placebo
Other: Dentifrice standard — Use of few of dentifrice on brushing for one week, twice day. It's for the positive control of fluoride
  Arms: Dentifrice standard; Placebo
Other: Dentifrice with tara gum — Use of few of dentifrice on brushing for one week, twice day. It's for analysis of negative control of fluoride and action only of tara gum.
  Arms: Dentifrice with tara gum; Placebo

SUMMARY:
The literature recognizes that fluoride is the most widely used and studied means for dental remineralization. The use of fluoride toothpaste in brushing is considered more rational method for the prevention of caries. However, the current challenge of toothpaste is the substantivity, so new compounds have been introduced into these formulations. This study aims to evaluate the in vivo effect of fluoride dentifrice containing a natural product - hydrocolloid tara gum - in fluoride retention in saliva and dental plaque. A study of the clinical and laboratory type, crossover, double-blind, randomized will be held. After sample calculation, the total of 12 individuals aged between 18 and 35 years old, healthy, decayed, missing, and filled teeth index less than 6 and residents in brazilian northeast capital will be part of the sample. Fluoride bioavailability will be evaluated in the biofilm and saliva after the use of fluoridated weekly. The biofilm will be assessed on 1h and 12 h after brushing; and unstimulated saliva in times of 3, 15, 30, 45, 60 minutes and 12 hours after. It will be 4 toothpastes: 1100ppm F- with hydrocolloid; F- 550ppm with hydrocolloid; 1100ppm F- without hydrocolloid; Without fluoride with hydrocolloid. Between weeks of use, brushing will be extended washout (without fluoride and no hydrocolloid) to avoid carryover effect. inferential data analysis will be carried out, considering the amount of alpha <0.05. So knowing that caries is a dynamic process, the largest fluoride retention in the oral fluids promoted by the hydrocolloid may have important impact on Des-Re process and in the control of dental caries.

DETAILED DESCRIPTION:
1. Study design It is a quantitative study of double-blind randomized crossover clinical type with inductive approach and documentation of technical and direct observation with measurements in the laboratory.

   In order to assess the bioavailability of intraoral fluoride week after the use of fluoride toothpastes containing natural hydrocolloid, it will be collected biofilm samples 1h and 12 h after brushing; and unstimulated saliva in times of 3, 15, 30, 45, 60 minutes and 12 hours after. The data will be obtained by physical and chemical analysis of the samples of fluoride (F). Therefore, the study will consist of two interrelated steps: a clinical phase for biofilm collection and saliva; and laboratory stage for fluoride analysis in the samples.

   Will be conducted pilot test with three participants before the start of the study.
2. Sample Size The sample size calculation was performed using fluoride concentration data in dental biofilm previous study and taking effect size difference between the experimental dentifrice (1100 ppm F with hydrocolloid) and positive control of at least 3.4 ppm of F- in biofilm after 12 hours, namely, 25%. Admitting experimental protocol with beta error of 10% alpha error of 5%, one-tailed and statistical power of 90%, the sample size was calculated for 6 people. For the calculation we used the Excel software and mathematical formula for clinical trials of superiority given. Adding sample loss resulted in 12 people.
3. Experimental Dentifrice For this study will be used five toothpastes: 1100ppm F- with hydrocolloid; F- 550ppm with hydrocolloid; 1100ppm F- without hydrocolloid; Without fluoride with hydrocolloid; Without fluoride and no hydrocolloid. The toothpaste, made available by the company from Brazil are packed in the same packaging and have the taste of tutti frutti. Except wash out the tubes with toothpaste will be identified by colors (yellow, green, red and blue) by an independent researcher. The color code will not be revealed to the participants nor the researcher who will accompany them. These will be drawn at random for daily use for seven days in four times, giving an interval of one week wash-out between them.

   In these periods of wash-out will use a toothpaste without fluoride and without hydrocolloid. In the end, all study participants will use the 5 experimental dentifrice at different times.
4. Clinical phase The participant will be informed about the study and after its acceptance, he/she will initiate the study. Initially will be clinical examination in order to report the presence of any of the exclusion criteria already listed. After verifying the absence of these criteria, there will be a dental prophylaxis pumice for removal of this biofilm and in some cases may be made supragingival scraping. The patient will be advised not to make use of any fluoride product during the experiment. At first, volunteers are instructed to use a toothpaste without fluoride and no hydrocolloid (wash out) the first week, in order to equate the study participants and eliminate any potential carryover effects of toothpaste used previously.

   The participant will get a tube of toothpaste and will be instructed to brush their teeth for 1 minute and rinse with 10 mL of water twice a day (morning and night). On the seventh day, the participant will be instructed to brush only the occlusal surfaces of your teeth, to allow biofilm accumulation of flat surfaces. When going to bed, you are warned not to eat or drink (except water) as well as not brushing your teeth until the next day. On the following morning, approximately 12 hours after the last brushing and fasting, the first dental biofilm sample and unstimulated saliva is collected. It will be used to remove biofilm Hollenback vestibular faces, interproximal, palatal and lingual right hemiarch and deposited in a pre-weighed Eppendorf tube in an analytical balance. To saliva collection, the participant, at rest, will be instructed to spit for a minute in a graduated glass tube. After that, the participant will brush the occlusal surfaces for 1 min and rinse with 10 mL of water. Soon after, will new collection of saliva and plaque. Saliva samples will give up in times of 3, 15, 30, 45 and 60 minutes after brushing, while the biofilm left hemiarch will be collected one hour after brushing. After the collection will be offered at breakfast organized by researchers participating in the crown of that research center.
5. Laboratorial phase Samples will be evaluated through physical-chemical analysis of fluoride using calibrated fluoride electrode. Samples will be analyzed for fluoride concentration using ion-specific electrode after diffusion facilitated with hexamethyl disiloxane (HMDS). The calibration curve is made for each analysis. All analyzes will be done in triplicate and be submitted for validation.
6. Data analysis The study data will be analyzed by inferential statistics considering p <0.05.

ELIGIBILITY:
Inclusion Criteria:

* resident in João Pessoa
* Decayed, Missing, Filled Index<6
* Healthy

Exclusion Criteria:

* orthodontic treatment
* gingivitis
* Periodontal disease
* Smokers
* Present active tooth decay
* Tooth sensitivity
* Those undergoing treatment with fluoride products and / or use of antimicrobials in the past four weeks

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Bioavailability of intraoral fluoride (biofilm and saliva) | six months

CONTACTS AND LOCATIONS:
Overall Officials: Fábio Sampaio, Doctor, Study Director — University Federal of Paraiba
Locations (1):
- Federal University of Paraíba, João Pessoa, Paraíba, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aguilar-Galvez A, Noratto G, Chambi F, Debaste F, Campos D. Potential of tara (Caesalpinia spinosa) gallotannins and hydrolysates as natural antibacterial compounds. Food Chem. 2014 Aug 1;156:301-4. doi: 10.1016/j.foodchem.2014.01.110. Epub 2014 Feb 6. PMID 24629972
- [Background] Buzalaf MA, Vilhena FV, Iano FG, Grizzo L, Pessan JP, Sampaio FC, Oliveira RC. The effect of different fluoride concentrations and pH of dentifrices on plaque and nail fluoride levels in young children. Caries Res. 2009;43(2):142-6. doi: 10.1159/000211717. Epub 2009 Apr 8. PMID 19365118
- [Background] Whitford GM, Wasdin JL, Schafer TE, Adair SM. Plaque fluoride concentrations are dependent on plaque calcium concentrations. Caries Res. 2002 Jul-Aug;36(4):256-65. doi: 10.1159/000063931. PMID 12218274
- [Background] Pessan JP, Silva SM, Lauris JR, Sampaio FC, Whitford GM, Buzalaf MA. Fluoride uptake by plaque from water and from dentifrice. J Dent Res. 2008 May;87(5):461-5. doi: 10.1177/154405910808700501. PMID 18434577
- [Background] Pessan JP, Pinto Alves KM, Italiani Fde M, Ramires I, Lauris JR, Whitford GM, Toumba KJ, Robinson C, Buzalaf MA. Distribution of fluoride and calcium in plaque biofilms after the use of conventional and low-fluoride dentifrices. Int J Paediatr Dent. 2014 Jul;24(4):293-302. doi: 10.1111/ipd.12073. PMID 25045768
- [Background] Pessan JP, Conceicao JM, Grizzo LT, Szekely M, Fazakas Z, Buzalaf MA. Intraoral fluoride levels after use of conventional and high-fluoride dentifrices. Clin Oral Investig. 2015 May;19(4):955-8. doi: 10.1007/s00784-015-1426-3. Epub 2015 Feb 14. PMID 25677244
- [Background] Duckworth RM, Jones S. On the relationship between the rate of salivary flow and salivary fluoride clearance. Caries Res. 2015;49(2):141-6. doi: 10.1159/000365949. Epub 2015 Jan 27. PMID 25634162
- [Background] Duckworth RM, Morgan SN, Gilbert RJ. Oral fluoride measurements for estimation of the anti-caries efficacy of fluoride treatments. J Dent Res. 1992 Apr;71 Spec No:836-40. doi: 10.1177/002203459207100S09. PMID 1592970
- [Derived] Alves VF, Moreira VG, Soares AF, de Albuquerque LS, Moura HS, de Oliveira Silva A, Sampaio FC. A randomized triple-blind crossover trial of a hydrocolloid-containing dentifrice as a controlled-release system for fluoride. Clin Oral Investig. 2018 Dec;22(9):3071-3077. doi: 10.1007/s00784-018-2395-0. Epub 2018 Feb 26. PMID 29484546